CLINICAL TRIAL: NCT03915912
Title: A Feasibility Study of Mindfulness Meditation Practice in Malignant Glioma Patients Throughout Standard of Care Chemoradiation
Brief Title: Mindfulness Meditation in Glioma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Duke Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00101218
Record Dates: First submitted 2019-04-12; First posted 2019-04-16 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Malignant Glioma
Keywords: Malignant Glioma; Mindfulness; Dina Randazzo; Meditation; Katherine Barnett Peters
MeSH Terms: conditions — Glioma | interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: Newly diagnosed malignant glioma patients will participate in six 1-hour mindfulness sessions over the phone, followed by one 1-hour in-person mindfulness session.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness meditation (Experimental): Newly diagnosed malignant glioma patients will participate in six 1-hour mindfulness sessions over the phone, followed by one 1-hour in-person mindfulness session. Patients will complete various Quality of Life questionnaires and distress measuring tools prior to initiating the mindfulness sessions, at the clinic visit following the mindfulness intervention, and ~2 months after completing the mindfulness intervention. Additionally, patients will be provided with supplemental materials including website references and guided audiotape meditations to guide their individual practice outside of the weekly guided sessions.
  Interventions: Behavioral: Mindfulness meditation

INTERVENTIONS:
Behavioral: Mindfulness meditation — The study intervention consists of seven mindfulness sessions (six 1-hour telephone sessions and one 1-hour in-person session). The six weekly telephone-based mindfulness sessions will occur in a one-on-one format and will be followed by one in-person, one-on-one session, which will occur at the post-chemoradiation standard of care clinic visit.

SUMMARY:
This pilot study is designed to determine the feasibility of providing a mindfulness meditation program to patients with newly diagnosed malignant glioma during standard of care chemoradiation. Newly diagnosed malignant glioma patients will participate in six 1-hour mindfulness sessions over the phone, followed by one 1-hour in-person mindfulness session. Patients will complete various Quality of Life questionnaires and distress measuring tools prior to initiating the mindfulness sessions, at the clinic visit following the mindfulness intervention, and ~2 months after completing the mindfulness intervention. Additionally, patients will be provided with supplemental materials including website references and guided audiotape meditations to guide their individual practice outside of the weekly guided sessions.

The main objective of this study is to assess the feasibility of a mindfulness meditation intervention program, designed to mitigate the distress associated with the disease and first line treatment of patients with malignant glioma, and to determine whether it merits additional research in a subsequent trial.

There are no risks associated with participation in this study.

DETAILED DESCRIPTION:
Fifteen newly diagnosed WHO grade III or IV malignant glioma patients will be enrolled to this pilot feasibility study. Following completion of informed consent, patients will complete a baseline assessment consisting of various QoL/distress assessments including the Trail Making Test, the Functional Assessment of Cancer Therapy-Cognitive Function (FACT-Cog), the Pittsburgh Sleep Quality Index (PSQI), the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F), the Functional Assessment of Cancer Therapy-Brain (FACT-Br), the Five Facet Mindfulness Questionnaire - short form (FFMQ-SF), the Functional Assessment of Chronic Illness Therapy-Spiritual Well-Being (FACIT-Sp12), the NCCN Distress Thermometer with Symptom Inventory, and the Hospital Anxiety and Depression Scale (HADS). They will then begin the mindfulness intervention, consisting of six weekly telephone-based mindfulness sessions followed by one in-person mindfulness session. Post-treatment measures and an Exit Survey will be administered following the one in-person mindfulness session. Two months later, the QoL, cognition and distress assessments will be repeated and a Final Exit Survey will be administered. The Exit Survey will ask the patient about their individual mindfulness practice during the intervention, their intention to continue the practice beyond participation in this study, their satisfaction with the services received, and their perception of the effectiveness of the program. The Final Exit Survey will ask the patient about their mindfulness practice since the Exit Survey, and their intention to continue with the mindfulness practice. The investigators will also collect demographic data such as age, marital status, education, employment, date of diagnosis and death, tumor grade, histology, and type of treatment from the patient.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age
2. NCCN distress scale ≥ 4 OR at least one of the following problems indicated on the NCCN distress thermometer worksheet: depression, fears, nervousness, sadness, worry, loss of interest in usual activities, sleep, memory, or fatigue
3. Karnofsky Performance Status (KPS) ≥ 70
4. Patient must have histologically confirmed, newly diagnosed WHO grade III or IV malignant glioma
5. Patient must be prior to a planned 6-week standard of care chemoradiation regimen
6. Patient can speak, read, and write English
7. Patient has access to a telephone for mindfulness training
8. Patient has access to internet

Exclusion Criteria:

1. Patients previously or currently practicing or participating in mindfulness meditation practice
2. Intermittent or active psychosis
3. Psychiatric hospitalization within the last 6 months
4. Hospitalized in a rehab facility within the last 6 months for substance abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2020-01-09 (Actual); Study Completion 2020-01-09 (Actual)

PRIMARY OUTCOMES:
Acceptability: Number of sessions that the patient attends | 6 weeks
  One measure of the acceptability of the mindfulness intervention is the number of sessions the patient attended. The number of patients who attend at least 3 of the 6 telephone-based mindfulness session in addition to the in-person session is reported.
Acceptability: Patients' satisfaction with the mindfulness sessions: The number of patients that respond either 'somewhat satisfied,' 'mostly satisfied,' or 'very satisfied' to the question 'How satisfied are you with the mindfulness sessions?' | 6 weeks
  One measure of the acceptability of the mindfulness intervention is the extent of satisfaction patients have with the mindfulness sessions. The number of patients that respond either 'somewhat satisfied,' 'mostly satisfied,' or 'very satisfied' to the question 'How satisfied are you with the mindfulness sessions?' on the exit survey is reported.
Acceptability: Percentage of patients who intend to continue meditation after study completion | 6 weeks
  One measure of the acceptability of the mindfulness intervention is the intent to continue practicing mindfulness meditation following study completion. The percentage of patients who respond 'yes' to the question 'Do you plan on continuing to practice mindfulness meditation?' on the 6-week exit survey is reported.
Acceptability: Percentage of patients who continued meditation practice during the 2 months after study completion | 4 months
  One measure of the acceptability of the mindfulness intervention is the percentage of patients that continued mindfulness meditation during the 2 months following the intervention as measured by question 'Did you continue your meditation practice after the training sessions?' captured on the final exit survey given 4 months after study initiation, which is 2 months after completing the mindfulness intervention. The percentage of patients responding 'yes' to this question is reported.
Demand: Total time required to enroll 15 patients | 2 years
  One measure of the demand of the mindfulness intervention is the length of time required to enroll 15 patients. The length of time in months needed to enroll 15 patients is reported.
Demand: Percentage of patients who enroll in the study | 2 years
  One measure of the demand of the mindfulness intervention is the percentage of patients enrolling in the study of those to which the study is offered. This percentage is reported.
Implementation: Percentage of patients who complete the study questionnaires | 4 months
  Implementation of the mindfulness intervention is measured by the percentage of patients who complete the study questionnaires measuring quality of life and evaluation of the mindfulness intervention at each time point of the study. Questionnaires are completed at baseline during screening, approximately 6 weeks post-baseline at the in-person mindfulness session, and 4 months post-baseline at the follow-up final exit survey. The percentage of patients who completed all questionnaires at each study time point is reported.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine B Peters, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Preston Robert Tisch Brain Tumor Center at Duke — https://tischbraintumorcenter.duke.edu/
- See also: Duke Cancer Institute — http://www.dukecancerinstitute.org/